CLINICAL TRIAL: NCT05960006
Title: An Observational Explorative Study to Determine Pharmacokinetic Changes of Ceftriaxone in Blood and Ascites in Patients Admitted With Decompensated Liver Cirrhosis With or Without Renal Impairment.
Brief Title: A Study to Determine Pharmacokinetic Changes of Ceftriaxone in Patients With Liver Cirrhosis
Acronym: TACTILE
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Marten A Lantinga, MD PhD, Consultant Hepatology, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W23_012 # 23.033
Record Dates: First submitted 2023-07-13; First posted 2023-07-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Antibiotic Toxicity; Liver Cirrhosis; Renal Insufficiency; Ceftriaxone Overdose; Ascites Hepatic; Infection, Bacterial
MeSH Terms: conditions — Liver Cirrhosis; Renal Insufficiency; Bacterial Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and ascites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- observational ceftriaxone: Patiënts with liver cirrhosis receiving ceftriaxone treatment.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — There are no risks associated with participation because only waste material (blood and ascites) will be used for analysis and no additional blood collection or paracentesis will be performed in addition to standard-of-care. Moreover, hospital admittance and discharge, indication for interventional procedures, indication/initiation/duration/dosing of ceftriaxone, indication/timing/frequency of blood withdrawal for standard of care biochemical analysis and microbiological culturing as the indication, timing, frequency and duration of paracentesis are all decided by the treating physician independent of participation in the study. There are no extra site visits nor extra days of hospital admission. There is no direct benefit for participants of this explorative study. .

SUMMARY:
The investigators designed an observational multicenter explorative in vivo study to investigate the changes in ceftriaxone pharmacokinetics in blood and ascites. The investigators will include a total of 20 patients with liver cirrhosis admitted to the ward of participating hospitals. Patients are eligible when receiving ceftriaxone and concomitantly receive paracentesis. The investigators will collect all available waste blood samples of each participant, starting from study entry up until 48 hours after the last dosing interval of ceftriaxone. The investigators will collect all available waste ascites samples of each participant up until 48 hours after the last dosing interval of ceftriaxone. Duration of the trial: The study duration is variable and depends on the duration of ceftriaxone treatment and duration of hospital admission, which both are determined by the treating physician and is not influenced by study participation. Patients will be eligible for study inclusion when patients received (a single dose of) ceftriaxone treatment and undergo paracentesis during ceftriaxone treatment. The study will end 48 hours after the last dosing interval of ceftriaxone or until hospital discharge, whichever comes first. Study timeline: The investigators expect to enrol 1-2 participants every month. The total enrolment time will thus be approximately 12 months.

DETAILED DESCRIPTION:
Objective: The primary objective is to determine the changes in ceftriaxone pharmacokinetics in blood and ascites in patients with decompensated liver cirrhosis to guide ceftriaxone dosing in these patients.

Study design: Observational explorative multicentre study

Study population: Adults (>18 years) with decompensated liver cirrhosis with the presence of ascites admitted to the clinical ward of participating centres who receive ceftriaxone and concomitantly undergo paracentesis during active antibiotic treatment.

Intervention: No intervention, the investigators will only collect the available waste blood and ascites samples.

Main study parameters/endpoints:

* Clearance (CL) of unbound ceftriaxone
* Volume of distribution (VD) of unbound ceftriaxone
* Penetration rate of unbound ceftriaxone from blood to ascites
* Elimination rate of unbound ceftriaxone from ascites by paracentesis

Secondary study parameters are:

* Target attainment of ceftriaxone in blood, defined as the unbound plasma concentration of ceftriaxone above at least one time the minimal inhibitory concentration (MIC) for 50% of the dosing interval (50%fT > 1MIC).
* Target attainment of ceftriaxone in ascites, defined as the unbound ascites concentration of ceftriaxone above at least one time the minimal inhibitory concentration (MIC) for 50% of the dosing interval (50%fT > 1MIC).
* Explorative analysis on the effects of liver disease severity (Child Pugh, MELD-score) and renal insufficiency (CKD-stage) on individual pharmacokinetic parameters

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical, radiological and/or histological diagnosis of liver cirrhosis and portal hypertension
* Presence of ascites
* Receiving ceftriaxone in the context of prophylaxis or treatment of infection
* Indication for diagnostic and/or therapeutic paracentesis
* Providing oral informed consent

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All admitted patients with the diagnosis of liver cirrhosis and ascites who receive at least a single dose of ceftriaxone during the current admission and receive diagnostic and/or therapeutic paracentesis following administration of ceftriaxone are suitable for inclusion in this study. The indication for diagnostic and/or therapeutic paracentesis is made upon the discretion of the treating physician following standard-of-care protocols.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Clearance (CL) of unbound ceftriaxone | 12 months
  Clearance (CL) of unbound ceftriaxone
Volume of distribution (VD) of unbound ceftriaxone | 12 months
  Volume of distribution (VD) of unbound ceftriaxone
Penetration rate of unbound ceftriaxone from blood to ascites | 12 months
  Penetration rate of unbound ceftriaxone from blood to ascites
Elimination rate of unbound ceftriaxone from ascites by paracentesis | 12 months
  Elimination rate of unbound ceftriaxone from ascites by paracentesis

SECONDARY OUTCOMES:
Target attainment of ceftriaxone in blood, defined as the unbound plasma concentration of ceftriaxone above at least one time the minimal inhibitory concentration (MIC) for 50% of the dosing interval (50%fT > 1MIC) | 12 months
  Target attainment of ceftriaxone in blood, defined as the unbound plasma concentration of ceftriaxone above at least one time the minimal inhibitory concentration (MIC) for 50% of the dosing interval (50%fT > 1MIC)
Target attainment of ceftriaxone in ascites, defined as the unbound ascites concentration of ceftriaxone above at least one time the minimal inhibitory concentration (MIC) for 50% of the dosing interval (50%fT > 1MIC) | 12 months
  Target attainment of ceftriaxone in ascites, defined as the unbound ascites concentration of ceftriaxone above at least one time the minimal inhibitory concentration (MIC) for 50% of the dosing interval (50%fT > 1MIC)
Explorative analysis on the effect of Child Pugh-score on individual pharmacokinetic parameters | 12 months
  Child Pugh score ranges from 5 points (minimum value) to 15 points (maximum value). Higher score means a worse outcome. Child Pugh score is a measure to determine the prognosis of patients with cirrhosis.
Explorative analysis on the effect of MELD-score on individual pharmacokinetic parameters | 12 months
  MELD-score (Model for End-Stage Liver Disease, version: original, pre-2016) ranges from 6 points (minimum value) to 40 points (maximum value). Higher score means a worse outcome. MELD-score quantifies end-stage liver disease for transplant planning.
Explorative analysis on the effect of CKD-stage on individual pharmacokinetic parameters | 12 months
  CKD (chronic kidney disease) stage ranges from stage 1 (minimum value) to stage 5 (maximum value). Higher score means a worse outcome. CKD-stage is based on the estimated glomerular filtration rate (eGFR, in mL/min/1.73m2) and refers to a measure of kidney function.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam university medical centers location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data is available upon reasonable request.